CLINICAL TRIAL: NCT05324943
Title: A Phase 1, Open-label, Safety, Tolerability, and Efficacy Study of FLT201 in Adult Patients With Gaucher Disease Type 1 (GALILEO-1)
Brief Title: A Gene Therapy Study in Patients With Gaucher Disease Type 1
Acronym: GALILEO-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spur Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLT201-01
Record Dates: First submitted 2022-02-28; First posted 2022-04-13 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Gaucher Disease, Type 1
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- FLT201 (Experimental): FLT201 is an advanced therapy investigational medicinal product (ATIMP) administered as a single intravenous infusion.
  Interventions: Genetic: FLT201

INTERVENTIONS:
Genetic: FLT201 — FLT201 is a replication-incompetent single-stranded (ss) recombinant adeno-associated virus (AAV) vector. The vector is composed of a ss DNA genome packaged in an AAV-derived protein capsid.

SUMMARY:
This study is a first-in-human, open-label, safety, tolerability, and efficacy study in adult patients with Gaucher disease Type 1. The aims are to investigate the safety/tolerability and efficacy of FLT201, and to investigate the relationship of FLT201 dose to augmentation of residual glucocerebrosidase (GCase) expression (activity and concentration), and its potential to improve the clinical phenotype by reduction and prevention of cellular accumulation of GCase substrate.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years of age.
2. Diagnosis of Gaucher disease Type 1 with deficient GCase enzyme activity ≤30% of normal in leukocytes at diagnosis.
3. All female patients of childbearing potential must not be lactating and must have a negative serum pregnancy test at screening and confirmed negative by urine testing prior to dosing on Day 1. Female patients of childbearing potential and male patients must be willing to follow protocol guidelines for barrier protection/contraception.
4. Able to give full informed consent for the trial.
5. Treatment status at screening (screening period is 16 weeks):

Treated with either enzyme replacement therapy (ERT) or substrate reduction therapy (SRT) and started this treatment at least 2 years prior to dosing with no change in regimen for the prior 3 months. ERT dose ≥15 U/kg and ≤60 U/kg every other week.

Exclusion Criteria:

1. Diagnosed or suspected Type 2 or Type 3 Gaucher disease (including any patient with eye movement abnormality on clinical examination).
2. Positive for neutralising antibodies to AAVS3 at screening.
3. Evidence of significant and persistent liver dysfunction at Screening defined as >1.5 x upper limit of normal (ULN) in alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin.
4. Evidence of any of the following at screening:

   1. Hb <8 g/dL.
   2. Platelets <45,000/mm3.
   3. Pulmonary hypertension.
   4. New osteonecrosis within 12 months of screening.
   5. Fragility fracture or bone crisis within 12 months of screening.
5. Hepatitis B surface antigen (HBsAg) positive at screening.
6. Hepatitis C antibody (Hep C Ab) positive and hepatitis C RNA polymerase chain reaction (PCR) (as follow-up test if Hep C Ab-positive)-positive at screening.
7. Cytomegalovirus (CMV) immunoglobulin G (IgG) and CMV DNA PCR-positive at screening.
8. Human immunodeficiency virus (HIV)-1 or -2 antibody positive at screening.
9. Patient has received live attenuated vaccination within 12 weeks prior to screening or intends to receive such vaccination during the study.
10. History of clinically-advanced liver disease e.g. cirrhosis, portal hypertension.
11. History of bone marrow transplant.
12. History of splenectomy (partial or total).
13. History of splenic infarct within 12 months of screening.
14. History of receiving any gene transfer medicinal product.
15. History of receiving any investigational therapy for Gaucher disease within 60 days of screening.
16. Participation in any other clinical study of an investigational medicinal product (IMP), and/or receiving any other IMP during the study.
17. History of idiopathic thrombocytopaenic purpura, thrombotic thrombocytopaenic purpura, thrombocytopaenia, anaemia, hepatomegaly, splenomegaly, and/or osteoporosis, unrelated to Gaucher disease.
18. History of, or active neoplastic disease within 5 years of screening (except for basal or squamous cell carcinoma of the skin or carcinoma in situ which has been definitively treated).
19. Subjects with uncontrolled cardiac failure, unstable angina, myocardial infarction, pulmonary hypertension or cardiac presentations including cardiac instability deemed significant by the investigator in the past 6 months
20. History of acute myocarditis or presence of acute myocarditis during screening.
21. History of substance abuse, including alcohol abuse or alcohol dependence.
22. Known or suspected intolerance, hypersensitivity or contraindication to the investigational medicinal product (IMP) and non-investigational medicinal products (NIMPs) or their excipients.
23. History of anaphylaxis or infusion related reactions to ERT.
24. Contraindication(s) to MRI. (e.g. ferromagnetic metallic implants, some types of pacing and defibrillator devices, nerve stimulators).
25. Any clinical condition (medical or psychiatric) that, in the opinion of the investigator, could jeopardise safety or compromise ability of the patient to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day 1 (dosing) through the final follow-up visit at Week 38
  Treatment-emergent adverse events (including dose-limiting toxicities), with AEs graded as mild/moderate/severe.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - Kaiser Permanente, Los Angeles, California
  - Lysosomal Rare Disorders Research and Treatment Center, Fairfax, Virginia
- Hospital de Clinicas de Porto Alegre (HCPA), Porto Alegre, Brazil
- SphinCS, Höchheim, Germany
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center - PPDS, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Hospital Quironsalud Zaragoza, Zaragoza, Spain
- United Kingdom (2):
  - Royal Free Hospital, London
  - Salford Royal Hospital, Salford